CLINICAL TRIAL: NCT01073540
Title: Prospective, Randomized, Open Label, Crossover Study to Compare the Bioavailability Between Optocef Suspension From Bayer (Cephalexin Suspension 250 mg/5 mL) and Equivalent Concentration of Keflex Pediatrico From Eli Lilly (Cephalexin Suspension 125 mg/5mL) in Healthy Subjects
Brief Title: Cross-over Study to Prove Bioequivalence Between Two Brands of Cefalexin Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Corporación Bonima S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14783
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Anti-Infective Agents
MeSH Terms: interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Cephalexin suspension (Optocef, BAYO5448)
- Arm 2 (Active Comparator)
  Interventions: Drug: Cephalexin suspension (Keflex)

INTERVENTIONS:
Drug: Cephalexin suspension (Optocef, BAYO5448) — Single dose of 500 mg / 10 mL
  Arms: Arm 1
Drug: Cephalexin suspension (Keflex) — Single dose of 500 mg / 20 mL
  Arms: Arm 2

SUMMARY:
A single dose, two treatments (two cephalexin suspension brands), two sequences, cross-over design was used with a washout of 7 days between the two study periods. Treatment groups balanced with the same number of healthy volunteers who were randomly (in two strata: male and female) assigned to the study drug administration sequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers age between 18 and 55 years old with normal vital signs, electrocardiogram (ECG), blood chemistry, liver function profile and urinalysis

Exclusion Criteria:

* History of illnesses or any organic abnormalities that could affect the results of the study
* History of tobacco or alcohol abuse or regular use of recreational or therapeutic drugs
* Subjects that have taken any medication within 14 days or that are in an elimination period of less than 7 half-lives (whichever is longest) before study startup

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Least square estimator of average maximum plasmatic concentration (log transformed) | After two months
Least square estimator of area under the pharmacokinetic curve (log transformed) | After two months

SECONDARY OUTCOMES:
Time at which maximum concentration is reached | After two months
Area under the pharmacokinetic curve from time=0 to last blood sample | After two months
Clearance constant of plasmatic concentration of study drug | After two months
Half life of plasmatic concentration of study drug | After two months
Adverse events collection | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Morelia, Michoacán, Mexico